CLINICAL TRIAL: NCT06355947
Title: Cycling Induced Motor Cortex Plasticity and Functional Improvement -the Dual Task Evaluation Model for Parkinson Disease
Brief Title: Cycling and Treadmill With Dual Task for Parkinson's Disease Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103-7445B
Record Dates: First submitted 2024-03-26; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease(PD)
Keywords: Gait; Cycling training; Treadmill training; Dual-task walking; Dual-task cycling
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Stage 1:Healthy people (No Intervention): To establish a baseline and ensure reliability, and to explore the relationship between dual-task gait performance and dual-task cycling
- No Intervention: Stage 2:PD people (No Intervention): To explore the relationship between dual-task gait and dual-task cycling performances in individuals with Parkinson's Disease (PD)
- Stage 3:PD cycling training group (Experimental): Cycling training conducted with cognitive tasks
  Interventions: Other: Cognitive cycling training
- Stage 3: PD treadmill training group (Experimental): Treadmill training conducted with cognitive tasks
  Interventions: Other: Cognitive treadmill training
- Stage 3:PD Control group (No Intervention): Control group

INTERVENTIONS:
Other: Cognitive cycling training — Cycling training conducted with cognitive tasks
  Arms: Stage 3:PD cycling training group
Other: Cognitive treadmill training — Treadmill training conducted with cognitive tasks
  Arms: Stage 3: PD treadmill training group

SUMMARY:
Motor impairment in lower extremities is common in individuals with Parkinson disease (PD). Development sensitive test for early motor deviations is important. Conventional walking test cannot induce the PD related motor impairments, such as freezing of gait. Therefore, finding a safe substitute test to induce PD related motor impairments is important.

Studies showed that working memory related dual task walking was a sensitive test for PD. However, the optimal cognitive test needs to be clarified. Studies also showed that the neuromuscular control mechanism of leg movements during cycling were similar to those during walking. Therefore, dual task cycling test is potential to be a safe and sensitive testing model.

Studies showed that exercise could improve cognitive function and induce brain plasticity. Dual task exercise training was shown to be more effective than single task exercise training for older people to prevent fall. Whether the added cognitive task could improve to detriment brain plasticity in PD should be investigated. Transcranial magnetic stimulation can evaluate the motor cortex plasticity on-invasively and can evaluate the exercise induced brain plasticity.

The purpose of this three-year project is to develop PD-sensitive. The purposes of the first year are to translate the dual task walking test to dual task cycling test, and to establish the reliability of the dual task cycling test.

The purposes of the second year are to compare the motor cortex plasticity induced by single task cycling versus dual task cycling and to compare the difference response between PD and healthy control people.

The purpose of the third year is to evaluate the effect of 8 week long term cycling training or treadmill training of individuals with PD on motor cortex plasticity, dual task performance, and ambulation ability.

ELIGIBILITY:
Health subjects:

Exclusion Criteria:

* Musculoskeletal injuries on legs.
* Osteoporosis.

PD subjects:

Inclusion Criteria:

- Clinical diagnosis of Parkinson disease.

Exclusion Criteria:

* Musculoskeletal injuries on legs
* Osteoporosis.
* Any peripheral or central nervous system injury or disease patients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Walking Speed | Baseline, 4 weeks and 8 weeks
  The time taken by participants to walk a standardized distance, typically expressed in centimeters per second (cm/s).
Step Length | Baseline, 4 weeks and 8 weeks
  The linear distance between the two ankles, typically expressed in centimeters(cm).
Step Time | Baseline, 4 weeks and 8 weeks
  The duration taken for one complete step, measuring from foot-off of one foot to the next foot-off of the same foot, usually expressed in seconds.
Power Spectral Density (PSD) | Baseline, 4 weeks and 8 weeks.
  Quantifies the power of EEG signals within specific frequency bands (e.g., delta, theta, alpha, beta, and gamma) over a period.
Task Accuracy | Baseline, 4 weeks and 8 weeks.
  The percentage of correct responses or actions made by participants in response to walking or cycling tasks.
Reaction Time | Baseline, 4 weeks and 8 weeks.
  The duration between the onset of task start time and the participant's response to it, typically expressed in second (s).
Balance Performance | Baseline, 4 weeks and 8 weeks
  Measured by the duration the stance can be maintained, typically expressed second.

SECONDARY OUTCOMES:
Double Support Time | Baseline, 4 weeks and 8 weeks
  The portion of the gait cycle where both feet are in contact with the ground, indicating the transition phase between steps, expressed as a percentage of the gait cycle or in seconds.
Single Support Time | Baseline, 4 weeks and 8 weeks
  The duration within the gait cycle when only one foot is in contact with the ground, typically measured in seconds or as a percentage of the total gait cycle.
Swing Time | Baseline, 4 weeks and 8 weeks
  The portion of the gait cycle where the foot is not in contact with the ground, moving forward to the next step. It is usually expressed as a percentage of the total gait cycle or in seconds.
Stance Time | Baseline, 4 weeks and 8 weeks
  The portion of the gait cycle when the foot is in contact with the ground, supporting body weight. It's typically expressed as a percentage of the total gait cycle or in seconds
Cadence | Baseline, 4 weeks and 8 weeks
  The number of steps an individual takes per minute, providing an overview of gait speed and rhythm, , expressed as steps per minute.
Heart rate | Baseline
  The number of heartbeats per minute on resting, walking or cycling tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan